CLINICAL TRIAL: NCT06838884
Title: An Alternative Assessment in Patients with Rheumatoid Arthritis: Comparing Bicycle Ergometer and 6 Minute Step Test and Proving the Validity of the 6 Minute Step Test
Brief Title: An Alternative Assessment in Patients with Rheumatoid Arthritis: 6 Minute Step Test
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Havvagül Doğan, Physiotherapy and Rehabilitation, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/15-25
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis (RA; 6 Minutes Stepper Test
Keywords: Rheumatoid arthritis; 6 minutes stepper test; Bicycle ergometer
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluated Group (Experimental): In this single-group study, two tests will be performed and compared. A 6-minute stepper test and a bicycle ergometer test will be applied.
  Interventions: Other: 6 minutes step test and bicycle ergometer

INTERVENTIONS:
Other: 6 minutes step test and bicycle ergometer — Evaluation

SUMMARY:
Although joint involvement is predominant, RA is a systemic disease that can affect many organs. RA is a disease that includes changes such as inflammation, joint pain, fatigue, increased risk of coronary and heart disease. In patients with RA, exercises should be planned for decreased muscle strength, endurance, aerobic capacity and affected normal joint movements. Aerobic exercise capacity should be measured for individualized exercise planning in rehabilitation. Bicycle ergometer, one of the aerobic capacity tests, has been used in rehabilitation for a long time. Although it is frequently used in rehabilitation, it has some disadvantages. Therefore, other tests such as the step test can be used to eliminate these disadvantages of the bicycle ergometer and to assess functional capacity. The 6-minute step test (6MST), which requires less time and space, can be used as an alternative to assess exercise capacity. Patients will be evaluated at Firat University Hospital. Patients diagnosed with RA, older than 18 years of age and with a body weight of 100 kg or less (maximum weight supported by the stepper) will be included in the study.

DETAILED DESCRIPTION:
Although joint involvement is predominant, RA is a systemic disease that can affect many organs. RA is a disease that includes changes such as inflammation, joint pain, fatigue, increased risk of coronary and heart disease. In patients with RA, exercises should be planned for decreased muscle strength, endurance, aerobic capacity and affected normal joint movements. Aerobic exercise capacity should be measured for individualized exercise planning in rehabilitation.The bicycle ergometer, which is one of the aerobic capacity tests, has been used in rehabilitation for a long time. Although it is frequently used in rehabilitation, it has some disadvantages. The bicycle ergometer may not always be consistent because it can vary depending on how fast the person is pedaling. It is also expensive equipment and may not be available in rehabilitation centers. In clinical settings, attention has been drawn to functional capacity tests, which can objectively assess exercise capacity, are easier to perform and do not require expensive equipment.Therefore, other tests such as the step test can be used to overcome these disadvantages of the bicycle ergometer and assess functional capacity. The 6-minute step test (6MST), which requires less time and space, can be used as an alternative to assess exercise capacity. Patients will be evaluated at Firat University Hospital. Patients diagnosed with RA, older than 18 years of age and with a body weight of 100 kg or less (maximum weight supported by the stepper) will be included in the study. Cosmed Fitmate Med, bicycle ergometer will be used. Before this test is performed, the patients' information will be entered into the device. Then a device that wraps around the patient's chest to measure HR values, a mask to measure VO2 values and a sphygmomanometer to measure blood pressure will be worn. The test will be done for as long as the patient can do it and will be finished at the patient's request. Post-test values will be recorded.

The patient will then be administered the 6MST test. This test will be performed according to the guidelines published by Borel et al. Before the test starts, the patient's heart rate, oxygen saturation, blood pressure, initial dyspnea and leg fatigue will be recorded. The stepper used can display the duration of the exercise, the number of steps per minute and the total number of steps. These values will be recorded after the test is finished. After the test, the patient's heart rate, oxygen saturation, blood pressure, dyspnea and leg fatigue will be recorded. The reliability of the 6 MST will then be decided by comparing these two test data.

ELIGIBILITY:
Inclusion Criteria:

* RA patient
* Over 18 years of age
* 100 kilos or less
* Patients who can walk independently without an assistive device

Exclusion Criteria:

* History of serious heart and lung disease
* Presence of severe musculoskeletal and joint disorders that may interfere with the conduct of the test
* Arthroplasty or major operations on knee and hip joints
* Uncontrolled hypertension
* Inability to participate in physical tests involving walking and cycling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-18 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Modified Borg Scale | up to 30 minutes
  The modified Borg scale is a validated scale for the subjective perception of dyspnea, used to verify the degree of respiratory distress. Exercise intensity is determined by individualized measurement. The 2002 guidelines of the American Thoracic Society recommend the modified Borg scale as an aid. This is a vertical scale measured from 0 to 10. Here 0 represents no symptoms and 10 represents maximum symptoms. In this study the modified Borg scale will be used to rate dyspnea and leg fatigue. The Borg scale will be printed out and this printout will be used for patient enumeration. The patient will be told what the numbers from 0 to 10 on the Borg scale mean. Instructions to the patient: "On the paper in your hand you see the numbers from 0 to 10. 0 means none, 10 means very severe. What the other numbers in between mean is written next to them. Now I want you to describe your breathing difficulty and leg fatigue with a number". After these instructions, the patient will be asked to n

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Merkez, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No